CLINICAL TRIAL: NCT04094337
Title: Implementing Internet-Assisted Treatment for Non-Cardiac Chest Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 815486
Record Dates: First submitted 2019-09-12; First posted 2019-09-18 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Chest Pain
Keywords: non-cardiac chest pain; NCCP; anxiety; internet-assisted treatment
MeSH Terms: conditions — Chest Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Eligible patients will be consecutively included and randomized to two groups, intervention group or control group. The investigators will use a web-based randomisation procedure, conducted at a place remote from where the study takes place.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-assisted treatment (Experimental): The intervention group will receive internet-assisted treatment comprising six web-based sessions, comprising information, exposure to physical activity, how worry can excess pain, physical reactions to pain and worry, consequences of avoidance, and specific panic treatment. The first session will be done at the hospital before discharge, the others at home. Between sessions there will be a brief telephone contact with a project worker.
  Interventions: Behavioral: Internet-assisted treatment
- Control group (No Intervention): The control group will receive treatment as usual, which is no specific treatment. The control group can however use the general health system as they like.

INTERVENTIONS:
Behavioral: Internet-assisted treatment — Internet-assisted treatment
  Arms: Internet-assisted treatment

SUMMARY:
This study aims to test Implementation of Internet-Assisted Treatment for Non-Cardiac Chest Pain at the Cardiac Department at Sørlandet Hospital. The internet-assisted treatment will be delivered by personnel working at the department. Effectiveness will be tested in an randomized controlled trial (RCT). The intervention has been tested in an RCT where the intervention was delivered by a cognitive behavioral therapy (CBT) specialist who also participated in developing the intervention. Presently the investigators will test if personnel working at the department, with minimal training in CBT, can deliver the intervention effectively.

DETAILED DESCRIPTION:
Most patients with chest pain referred to hospital do not have a cardiac illness. Non-cardiac chest pain (NCCP) is often followed by persistent distress and reduced quality of life, and societal costs are nearly equal to those of cardiac patients. Research suggests that face-to-face CBT is effective, but this has not been implemented as standard treatment. The investigators plan to test an easily implementable internet-assisted treatment for NCCP patients delivered by personnel already working at the department.

Patients will be recruited at the chest pain unit at Sørlandet Hospital, Kristiansand, and will be recruited after they have finished their cardiac examination.

The intervention group will receive six web-based sessions, comprising information, exposure to physical activity, how worry can excess pain, physical reactions to pain and worry, consequences of avoidance, and specific panic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Non-Cardiac Chest Pain

Exclusion Criteria:

* Language difficulties
* Unable to perform at least moderate physical activity due to physical constraints
* Obvious cognitive impairment (e.g mentally retarded, psychotic, dementia or intoxicated)
* no regular access to a computer/tablet computer with internet connection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 169 (Estimated)
Dates: Start 2019-10-26 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Body Sensations Questionnaire (BSQ) | 58 weeks
  BSQ is an 17-item self-report-questionnaire which measures fear of different bodily sensations. Each item is rated on a five-point Likert scale ranging from 1 to 5. Total range 17-85 where higher score represents more symptoms. Primary outcome is difference in mean score between intervention arm and control arm for BSQ at end of treatment (6 weeks after randomization for both arms). Difference in mean scores between arms will also be assessed at pretreatment/baseline, and at 3 months and 12 months after end of treatment (18 weeks and 58 weeks after randomization). There is no predefined clinical relevant effect for this measure. The investigators will use a distribution based method. Clinical relevant effect is defined as improvement of more than 0.5 standard deviation compared to baseline.

SECONDARY OUTCOMES:
Change in Cardiac Anxiety Questionnaire (CAQ) | 58 weeks
  CAQ is an 18-item self-report-questionnaire which measures hearth related anxiety/fear, attention, avoidance and safety seeking behavior. Each item is rated on a five-point Likert scale ranging from 0 to 4. Total range 0-72 where higher score represents more symptoms. Primary outcome is difference in mean score between intervention arm and control arm for CAQ at end of treatment (6 weeks after randomization for both arms). Difference in mean scores between arms will also be assessed at pretreatment/baseline, and at 3 months and 12 months after end of treatment (18 weeks and 58 weeks after randomization). There is no predefined clinical relevant effect for this measure. The investigators will use a distribution based method. Clinical relevant effect is defined as improvement of more than 0.5 standard deviation compared to baseline.
Change in Brief Illness Perception Questionnaire (BIPQ) | 58 weeks
  BIPQ is an 8-item self-report-questionnaire which assess the patient's perception/beliefs about their symptoms. Each item is rated on a 0-10 scale. The items represent different components/dimensions. Secondary outcome is difference in mean score between intervention arm and control arm for item 1, 5, 6 and 8 at end of treatment (6 weeks after randomization for both arms). Difference in mean scores between arms will also be assessed for item 1, 5, 6 and 8 at pretreatment/baseline, and at 3 months and 12 months after end of treatment (18 weeks and 58 weeks after randomization). There is no predefined clinical relevant effect for this measure. The investigators will use a distribution based method. Clinical relevant effect is defined as improvement of more than 0.5 standard deviation compared to baseline.
Change in Patient Health Questionnaire (PHQ-9) | 58 weeks
  PHQ-9 is an 9 item self-report-questionnaire which assess depression symptoms. Each item is rated on a 0-3 scale. Total range 0-27 where higher score represents more symptoms. Secondary outcome is difference in mean score between intervention arm and control arm for PHQ-9 at end of treatment (6 weeks after randomization for both arms). Difference in mean scores between arms will also be assessed at pretreatment/baseline, and at 3 months and 12 months after end of treatment (18 weeks and 58 weeks after randomization).
Change in EQ-5D-5L | 58 weeks
  EQ-5D-5L is an 5 item (plus a visual analog scale) self-report-questionnaire assessing health related quality of life. Secondary outcome is difference in mean score between intervention arm and control arm for EQ-5D-5L at end of treatment (6 weeks after randomization for both arms). Difference in mean scores between arms will also be assessed at pretreatment/baseline, and at 3 months and 12 months after end of treatment (18 weeks and 58 weeks after randomization). Distribution based methods are commonly used, defining improvement of 0.2 or 0.5 standard deviation as clinical relevant. The investigators define a minimal clinical relevant improvement to be 0.2 standard deviation in EQ-5D-5L.
Change in self-developed questions | 58 weeks
  Questions regarding:
  1. Impact on social, work and Family life
  2. Frequency of chest pain
  3. Avoidance of physical activity due to chest pain
  4. Physical activity level

OTHER OUTCOMES:
PHQ-9 | 58 weeks
  Total range of PHQ-9 is 0-27. A score of 5 or above is defined as cut-off for mild depressive symptoms. The investigators will sub-group participants with a prescore of 5 or above on PHQ-9 to evaluate if this subgroup has:
  1. Effect of the intervention on the primary/secondary measures and how this compares to the Whole Group
  2. Evaluate if a score of 5 or above can predict outcome for these patients

CONTACTS AND LOCATIONS:
Overall Officials: Frode Gallefoss, PhD, Study Director — Head of Clinical Research; Egil Jonsbu, PhD, Principal Investigator — Researcher
Locations (1):
- Sorlandet Sykehus HF, Kristiansand, Vest-Agder, Norway

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 12 months of study completion.
Access Criteria: Data Access requests will be reviewed by the science unit at Sørlandet Hospital, Norway. Requestors will be required to sign a Data Access Agreement.